CLINICAL TRIAL: NCT03376217
Title: Assessing the Effectiveness of Community Delivery of Intermittent Preventive Treatment in Pregnancy (IPTp) in Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kamuzu University of Health Sciences (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Ministry of Health, Malawi (Other Government); Peace Corps (Other); Management Sciences for Health (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Julie Gutman, Medical epidemiologist, Kamuzu University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P.08/17/2232
Record Dates: First submitted 2017-12-06; First posted 2017-12-18 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Malaria in Pregnancy
Keywords: malaria; malaria in pregnancy; intermittent preventive treatment in pregnancy (IPTp); community health workers; Sulfadoxine-pyrimethamine (SP)
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): IPTp delivered at antenatal clinic
- Intervention (Experimental): IPTp delivered by HSAs
  Interventions: Other: IPTp delivered by HSAs

INTERVENTIONS:
Other: IPTp delivered by HSAs — Pregnant women will have the option to receive IPTp-SP from Health surveillance assistants (HSAs). SP is recommended in Malawi for prevention of malaria during pregnancy, but currently it is only available at antenatal clinics.
  Other Names: community IPTp (cIPTp)
  Arms: Intervention

SUMMARY:
The overall aim of the study is to learn whether utilization of Health Surveillance Assistants (HSAs) for delivery of intermittent preventive treatment of malaria in pregnant women (IPTp) can increase coverage of three or more IPTp doses compared to IPTp delivery only at antenatal clinics (ANC), while at the same time improve or maintain ANC attendance. This will be a cluster randomized trial, including a total of 20 health facilities (HF) which will be randomly assigned to either the intervention (10) or non-intervention group (10); all HSAs affiliated with a HF will be in the same group.

DETAILED DESCRIPTION:
Project Background WHO recommends the use of intermittent preventive treatment in pregnancy (IPTp) with sulfadoxine-pyrimethamine (SP) to prevent the adverse effects of malaria in pregnancy. In 2012, in an effort to boost uptake, the World Health Organization (WHO) updated its policy promoting initiation of IPTp-SP as early as possible during the second trimester and at every scheduled antenatal clinic (ANC) visit thereafter, as long as the visits were at least one month apart. Despite this recommendation, progress has been slow, and no sub-Saharan African country has achieved the 85% coverage target set by the President's Malaria Initiative (PMI). Malawi was the first country to adopt IPTp-SP, and though it had early gains, these have remained stagnant. Coverage of 2 doses of IPTp-SP was 42.9% in 2004 (DHS), 53.8% in 2010 (DHS), and remained only 63% as of 2014 (MIS), despite the fact that >95% of women make 2 or more visits to the ANC, with 44% making four or more visits, and despite the fact that the median gestational age at the first visit is 5.6 months. Clearly, a novel approach to ensure earlier presentation at ANC and increase IPTp delivery is needed to boost coverage to the 85% target. Community delivery of IPTp has been suggested as a means to improve coverage, however, there is concern that this could also lead to reduced antenatal care (ANC) visits. Thus, it is relevant to assess whether there is a benefit of community delivery of IPTp-SP under the current policy advocating IPTp at each ANC visit, whether this approach is feasible, both from the standpoint of service delivery as well as data collection, and ensure that there is no adverse effect on ANC attendance prior to large scale roll-out.

Study Aims Broad objective: The overall aim of the study is to learn whether utilization of Health Surveillance Assistants (HSAs) for delivery of intermittent preventive treatment of malaria in pregnant women (IPTp) can increase coverage of three or more IPTp doses compared to IPTp delivery only at antenatal clinics (ANC), while at the same time improve or maintain ANC attendance

Specific objectives Primary objective

1. Determine the effect of community-based IPTp delivery by HSAs compared with facility-based IPTp delivery on IPTp coverage (including 1, 2, 3, and 4 doses) and ANC coverage (including 1, 2, 3, and 4 visits) Secondary objectives
2. Document the level of service delivery by HSAs
3. Assess women's knowledge of HSAs and attitudes about receiving IPTp from a HSA
4. Assess the feasibility of scaling-up community delivery of IPTp from the perspective of health facility staff, and HSAs..
5. Assess the acceptability of community delivery of IPTp from health facility staff, HSAs, and women.
6. Assess the factors which may affect the scale-up of community delivery of IPTp from the perspective of health facility staff, HSAs, and women.
7. Assess incremental costs of community-based IPTp delivery compared to HF based IPTp delivery from both provider and household perspectives.

Methodology Study design: This will be a cluster randomized trial, including a total of 20 health facilities (HF) which will be randomly assigned to either the intervention (10) or non-intervention group (10); all HSAs affiliated with a HF will be in the same group.

The study will use baseline and end line cross sectional household surveys, midline and post-intervention in-depth interviews with health facility staff and HSAs, pre- and post-intervention in-depth interviews with women, and focus group discussions with HSAs to achieve the objectives.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women:

* All pregnant women residing in study catchment area are eligible to receive SP from HSAs, with the exception of HIV positive women.
* To be included in the women's question portion of the baseline and end line household surveys, women must be between the ages of 16-49 years, have been pregnant/delivered in the previous 12 months, consent to participation, and will be eligible for inclusion in surveys regardless of where the woman gave birth (i.e., whether at home or in facility). All pregnant/recently pregnant women will be included in the cross sectional survey, but the sample size is calculated in order to identify those who have completed pregnancies in the past 12 months. There were be a very short subset of demographic and knowledge questions which will be asked of all households during the baseline and end line surveys, regardless of whether there are any recently pregnant women in the household.

Providers:

* At each facility we will randomly select one ANC provider who has had at least six months of work experience
* HSA supervisor
* Health facility in-charge

HSAs:

• All HSAs working in the study areas will be eligible; we will select at least 36 at random to be participate in interviews and focus groups discussions.

Exclusion Criteria:

Pregnant women: Women who experienced a delivery in the past 12 months, but are <16 or >49 years will be excluded. Those who last delivered a child over twelve months ago will be excluded from survey questions specific to recently pregnant women, but may answer questions related to community perception or general demographics. For qualitative research, the same criteria will be used.

Health facility providers: Those who have been working in the health service for less than six months will not be interviewed due to low levels of relevant experience or exposure to the intervention.

HSAs: All HSAs are eligible to participate.

Ages: 16 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1447 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
3 or more doses of IPTp (IPTp3+) | through study completion, 18 months
  Proportion of recently pregnant women who received at least 3 doses of IPTp

SECONDARY OUTCOMES:
IPTp doses received | through study completion, 18 months
  Proportion of women who received 1, 2, or 4 or more dose of IPT
IPTp doses delivered by ANC | through study completion, 18 months
  Proportion of doses delivered by the HSA vs at the ANC
Total ANC visits | through study completion, 18 months
  proportion of women who made 1, 2, 3, 4, or more ANC visits
Gestational age at first IPTp | through study completion, 18 months
  gestational age at the time of first ANC and at 1st dose of IPTp

CONTACTS AND LOCATIONS:
Overall Officials: Jobiba Chinkhumba, MBBS PhD, Principal Investigator — Malaria Alert Center, Malawi College of Medicine; Julie Gutman, MD MSc, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Malaria Alert Center, University of Malawi College of Medicine, Liwonde, Malawi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Okeibunor JC, Orji BC, Brieger W, Ishola G, Otolorin E', Rawlins B, Ndekhedehe EU, Onyeneho N, Fink G. Preventing malaria in pregnancy through community-directed interventions: evidence from Akwa Ibom State, Nigeria. Malar J. 2011 Aug 5;10:227. doi: 10.1186/1475-2875-10-227. PMID 21819579
- [Background] Ndyomugyenyi R, Tukesiga E, Katamanywa J. Intermittent preventive treatment of malaria in pregnancy (IPTp): participation of community-directed distributors of ivermectin for onchocerciasis improves IPTp access in Ugandan rural communities. Trans R Soc Trop Med Hyg. 2009 Dec;103(12):1221-8. doi: 10.1016/j.trstmh.2009.03.006. Epub 2009 May 20. PMID 19467686
- [Background] Mbonye AK, Magnussen P, Bygbjerg IB. Intermittent preventive treatment of malaria in pregnancy: the effect of new delivery approaches on access and compliance rates in Uganda. Trop Med Int Health. 2007 Apr;12(4):519-31. doi: 10.1111/j.1365-3156.2007.01819.x. PMID 17445143
- [Background] Msyamboza KP, Savage EJ, Kazembe PN, Gies S, Kalanda G, D'Alessandro U, Brabin BJ. Community-based distribution of sulfadoxine-pyrimethamine for intermittent preventive treatment of malaria during pregnancy improved coverage but reduced antenatal attendance in southern Malawi. Trop Med Int Health. 2009 Feb;14(2):183-9. doi: 10.1111/j.1365-3156.2008.02197.x. Epub 2009 Jan 15. PMID 19207178
- [Background] Gies S, Coulibaly SO, Ky C, Ouattara FT, Brabin BJ, D'Alessandro U. Community-based promotional campaign to improve uptake of intermittent preventive antimalarial treatment in pregnancy in Burkina Faso. Am J Trop Med Hyg. 2009 Mar;80(3):460-9. PMID 19270299
- [Derived] Rubenstein BL, Chinkhumba J, Chilima E, Kwizombe C, Malpass A, Cash S, Wright K, Troell P, Nsona H, Kachale F, Ali D, Kaunda E, Lankhulani S, Kayange M, Mathanga DP, Munthali J, Gutman JR. A cluster randomized trial of delivery of intermittent preventive treatment of malaria in pregnancy at the community level in Malawi. Malar J. 2022 Jun 21;21(1):195. doi: 10.1186/s12936-022-04216-4. PMID 35729612